CLINICAL TRIAL: NCT05012592
Title: Reducing Malnutrition and Helminthic Infectious Disease Among Primary School Children
Brief Title: Reducing Malnutrition and Helminthic Infectious Disease Among Primary School Children by the School Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: North South University (Other)
Responsible Party: Principal Investigator, Sadia Aivey, Principal Investigator, Hiroshima University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/OR-NSU/IRB/0701; 21H03250 (Other Grant/Funding Number: Japan Society for the Promotion of Science (JSPS))
Record Dates: First submitted 2021-08-11; First posted 2021-08-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Malnutrition, Child; Intestinal Worms
Keywords: Malnutrition; Intestinal worm infestation; School nurse; Primary school children
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Health assessment (health checkup) and health awareness program to reduce malnutrition and helminth infestation among primary school children
  Interventions: Behavioral: Health Awareness Program TO Reduce Malnutrition and Helminth Infestation among Primary School children
- Comparison group (No Intervention): Health assessment (health checkup) was provided but no health educational intervention during the intervention period

INTERVENTIONS:
Behavioral: Health Awareness Program TO Reduce Malnutrition and Helminth Infestation among Primary School children — This interventional study period started from September 2021 up to September 2022 (13 months) by school nurses to implement HAPSC. After completing four to five months of the educational session the school nurse will collect midline follow-up data and the endline data will be collected at the end of the interventional study. In this period a total of nine months (except annual leave) will be considered an interventional education period. The intervention group will receive one educational session per week every month. School nurses will be assigned for each class to provide health education. Each session will be conducted for a maximum of 45 minutes. The community worker will be assigned to assist the school nurse and they will communicate with the child's parents about their child's healthy nutrition and good hygiene practice. The significance of healthy eating and hygiene behavior for the children will be shared with the child's parents or guardians properly.
  Arms: Intervention Group

SUMMARY:
Title: Reducing malnutrition and helminthic infectious disease among primary school children by the school nurses: School-based non-randomized study in a developing country

Introduction: Globally, malnutrition alone with the infectious disease a widespread problem among primary school (5 to 12 years) children. Infectious diseases such as worm infestations are aggravated with nutritional disorders which most often lead to anemia and several complications. The prevalence of malnutrition and intestinal worm infestation/ helminthic infection is still high and the awareness level of those issues is immensely poor. However, there are limited studies that evaluated the impact of increasing health awareness by the development of the Health Awareness Program for Primary School Children (HAPSC) which is conducted by the experimentally placed school nurse in Bangladesh.

Objective: To increase health awareness and knowledge towards reducing malnutrition and intestinal worm infestation by implement and evaluate the impact of the Health Awareness Program for Primary School children (HAPSC) in Bangladesh.

Methods:

Design: A prospective, open-label, parallel-group (1:1), cluster non-randomization controlled trial (NRCT)

Site and sample: School children from four primary schools in the rural areas of North Matlab at Chandpur district at Chittagong division in Bangladesh.

Duration: The duration of this study is from August 2021 to March 2024 (32nd months).

Outcome variables:

Primary: changes in malnutrition among primary school children. Secondary: Evaluate and reduce the prevalence of intestinal worm infestation, increase awareness and knowledge regarding malnutritional and intestinal worm infestation, improvement of health behavior (eating and hygiene), frequency of school absent days, and health-related quality of life.

Conclusion: Health education by the health professional in the school setting may be an effective method for improving health behavior, and increasing awareness and knowledge levels about malnutrition and intestinal worm infestation from early childhood.

ELIGIBILITY:
Inclusion Criteria:

* The primary school children who are studying in class 1 to class 5 among male, female or others gender.
* The children's parents or legal guardians would like to give consent and are willing to participate in the study.
* Those, who will be agreed to receive health check-ups, answer questionnaires and are willing to give the sample for laboratory investigation.
* Who will stay in the same school and area till study completion.

Exclusion Criteria:

* The child is absent from school during the health checkup periods (at baseline) due to severe illness or without any reason and information.
* Who does not want to give consent and is not willing to participate.
* Who does not want to share their information and does not want to give the sample for laboratory investigations.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 604 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in malnutrition rate among primary school children | Baseline, 4th/ 5th month after baseline (Midline) and 12th month after baseline (Endline)
  The primary outcome will be evaluated by anthropometric health assessment (Body mass index).
  To calculate BMI, the body weight and height will be used following the BMI formula (BMI = weight (kg) / (height)^2 (m)^2) provided by World Health Organization (WHO). Children's nutritional status and BMI-for-age will be measured by comparing the z- scores against the WHO growth reference 2007 tables for 5-19 years. The cut-off values for overweight and obesity are > + 1SD, > + 2SD respectively. On the other hand, the cut-off value for thinness is <- 2SD>.

SECONDARY OUTCOMES:
Change of the prevalence of intestinal worm infestation among primary school children | Baseline and 12th month after baseline (Endline)
  Evaluate by health assessment and laboratory test for helminth ova and the parasite
Change of the children's eating and drinking behavior, and health-related hygiene behavior | Baseline, 4th/ 5th month after baseline (Midline) and 12th month after baseline (Endline)
  Evaluate by using a questionnaire which is developed by the researcher
Change of the awareness and knowledge regarding malnutrition and intestinal worm infestation | Baseline, 4th/ 5th month after baseline (Midline) and 12th month after baseline (Endline)
  Evaluate by using a questionnaire which is developed by the researcher
Change of the frequency and number of school absent days among the children | Baseline, 4th/ 5th month after baseline (Midline) and 12th month after baseline (Endline)
  Evaluate by using a questionnaire which is developed by the researcher
Measuring the changes of Health-related quality of life (HRQoL) of the children | Baseline, 4th/ 5th month after baseline (Midline) and 12th month after baseline (Endline)
  Evaluate by using KIDSCREEN survey form, parents' version

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Aivey, Principal Investigator — Hiroshima University
Locations (1):
- North South University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
When the data will be available and we will share the data according to the recommendations of the clinical trial registration and the requests of the journals.